CLINICAL TRIAL: NCT03033303
Title: Hu3F8/GM-CSF Immunotherapy Plus Isotretinoin for Consolidation of First Remission of Patients With High-Risk Neuroblastoma: A Phase II Study
Brief Title: A Study of the Effect of Hu3F8/GM-CSF Immunotherapy Plus Isotretinoin in Patients in First Remission of High-Risk Neuroblastoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Y-mAbs Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 16-1643
Record Dates: First submitted 2017-01-24; First posted 2017-01-26 (Estimated); Last update posted 2025-10-07 (Actual); Status verified 2025-09

CONDITIONS: Neuroblastoma
Keywords: Hu3F8; GM-CSF; Isotretinoin; 16-1643
MeSH Terms: conditions — Neuroblastoma | interventions — naxitamab; Granulocyte-Macrophage Colony-Stimulating Factor; Isotretinoin

STUDY DESIGN:
Intervention Model Description: In this phase II single arm trial, patients with HR-NB in first CR or VGPR undergo consolidation by using hu3F8/GM-CSF.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Hu3F8/GM-CSF Plus Isotretinoin (Experimental): In this phase II single arm trial, patients with HR-NB in first CR or VGPR undergo consolidation by using hu3F8/GM-CSF x5 cycles and isotretinoin x6 cycles. Isotretinoin starts after cycle 2 of hu3F8/GM-CSF.
  Interventions: Biological: Hu3F8; Drug: GM-CSF; Drug: Isotretinoin

INTERVENTIONS:
Biological: Hu3F8 — Day 1: hu3F8 infused iv over ~30 to 90 minutes. Day 3: hu3F8 infused iv over ~30 to 90 minutes. Day 5: hu3F8 infused iv over ~30 to 90 minutes.
Drug: GM-CSF — Days -4 to 0: GM-CSF 250 mcg/m2/day, subcutaneously. Days 1 to 5: GM-CSF 500 mcg/m2/day, subcutaneously.
Drug: Isotretinoin — Isotretinoin is administered at 160 mg/m2/d, divided into two doses, x14 days.

SUMMARY:
The purpose of this study is to test see the combined effects of the study drug called Humanized 3F8 (Hu3F8) when used with granulocyte-macrophage colony stimulating factor (GM-CSF). Hu3F8 plus GM-CSF could prevent your neuroblastoma from growing, but it could also cause side effects.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of NB as defined by a) histopathology (confirmed by the MSK Department of Pathology), or b) BM metastases or MIBG-avid lesion(s) plus high urine catecholamine levels.
* Patients must have high-risk NB (MYCN-amplified stage 2/3/4/4S of any age and MYCN-nonamplified stage 4 in patients greater than 18 months of age).
* Patients must be in first CR/VGPR
* Patients must have a negative human anti-hu3F8 antibody (HAHA) titer

Exclusion Criteria:

* Existing major organ dysfunction, i.e., renal., cardiac, hepatic, neurologic, pulmonary, or gastrointestinal toxicity ≥ grade 3, with the exception of hearing loss and hematologic toxicity.
* Active life-threatening infection.
* Inability to comply with protocol requirements

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2017-01-23 (Actual); Primary Completion 2025-09-29 (Actual); Study Completion 2025-09-29 (Actual)

PRIMARY OUTCOMES:
relapse-free survival (RFS) | 2 years
  Patients are considered a response failure under this protocol if progressive disease is evident before two years. Deaths from toxicity attributable to protocol treatment will be counted as events. Patients who withdraw or are lost to followup before two years will be considered as progressions.

CONTACTS AND LOCATIONS:
Overall Officials: Brian H. Kushner, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kushner BH, Modak S, Mauguen A, Basu EM, Kramer K, Roberts SS, Cheung IY, Cheung NV. A Phase II Trial of Naxitamab plus Stepped-up Dosing of GM-CSF for Patients with High-Risk Neuroblastoma in First Complete Remission. Clin Cancer Res. 2025 May 15;31(10):1877-1884. doi: 10.1158/1078-0432.CCR-24-3427. PMID 40067131
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm